CLINICAL TRIAL: NCT02691884
Title: The Effect of Pressure Exerted on the Maternal Abdominal Wall by the Ultrasound Probe on Fetal Heart Rate
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0149-14-MMC
Record Dates: First submitted 2016-02-21; First posted 2016-02-25 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-02

CONDITIONS: Pregnancy
Keywords: Heart Rate, Fetal; Electronic Fetal Monitoring; Transducers, Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients before/after Pressure Exertion: 100 pregnant patients at term in low risk pregnancies, undergoing a routine cardiotocography, will experience different amounts of manual pressure on their abdomen. The amount of pressure applied will be recorded and the fetal heart rate will be compared before and at the time of maternal abdominal pressure.
  Interventions: Procedure: maternal abdominal pressure

INTERVENTIONS:
Procedure: maternal abdominal pressure — The fetal cardiac response of either acceleration, deceleration or no change at all to the fetal heart- will be recorded and later on analyzed in reference to the amount of pressure applied from the 20th minute of CTG and for 5 minutes, using the FSR 400 sensor.

SUMMARY:
The aim of the study is to assess the change of fetal heart rate in response to the amount of pressure exerted on the maternal abdomen. The amount of pressure will be quantified using an electronic pressure sensor (FSR 400- Round Force Sensor, Interlink).

DETAILED DESCRIPTION:
Previous studies have shown a fetal cardiovascular effect to the pressure exerted on the maternal abdomen. Our null hypothesis is that there is a correlation between fetal heart rate changes and pressure exerted on the fetus through the maternal abdomen.

Women at term pregnancy coming for a routine cardiotocography monitor, will undergo 5 minutes of quantified pressure on their abdomen, using the electronic pressure sensor. The amount of pressure will be recorded as well as the fetal heartbeat baseline and changes to the heart rate following the application of pressure.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* singleton pregnancy
* term (37-41 weeks of gestation)
* consented
* undergoing routine cardiotocography (CTG)

Exclusion Criteria:

* referred to the ER due to non reassuring fetal heart rate (NRFHR)
* recognition of NRFHR pattern on CTG at the ER
* self reporting of reduced fetal movement perception
* unconsented patient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Term singleton pregnancies in patients over 18 years of age, undergoing routine CTG for various indications- growth monitoring, gestational diabetes monitoring, post term, etc.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-01 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Changes in fetal baseline heart rate, including accelerations and decelerations | immediately after applying pressure to the maternal abdomen
  pressure will be applied after the 20th minute of CTG monitoring and for a total of 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Tal Weissbach, MD, Principal Investigator — Meir Medical Center, Tel Aviv University
Locations (1):
- Meir Medical Center, Kefar Sava, Israel

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Ramon y Cajal CL. Umbilical vein and middle cerebral artery blood flow response to partial occlusion by external compression of the umbilical vein (pressure test). J Matern Fetal Neonatal Med. 2002 Aug;12(2):104-11. doi: 10.1080/jmf.12.2.104.111. PMID 12420840
- [Result] Su YM, Lv GR, Chen XK, Li SH, Lin HT. Ultrasound probe pressure but not maternal Valsalva maneuver alters Doppler parameters during fetal middle cerebral artery Doppler ultrasonography. Prenat Diagn. 2010 Dec;30(12-13):1192-7. doi: 10.1002/pd.2648. PMID 21064194
- [Result] Vyas S, Campbell S, Bower S, Nicolaides KH. Maternal abdominal pressure alters fetal cerebral blood flow. Br J Obstet Gynaecol. 1990 Aug;97(8):740-2. doi: 10.1111/j.1471-0528.1990.tb16250.x. No abstract available. PMID 2205291
- [Result] Alpert Y, Ben-Moshe B, Shvalb N, Piura E, Tepper R. The Effect of the Pressure Exerted on the Maternal Abdominal Wall by the US Probe on Fetal MCA Peak Systolic Velocity. Ultraschall Med. 2017 Jan;38(1):44-50. doi: 10.1055/s-0035-1553332. Epub 2015 Sep 30. PMID 26422667